CLINICAL TRIAL: NCT06443996
Title: Effects of Sleep Quality and Mental Status on Early Postoperative Recurrence and Prognosis in Patients With Colorectal Cancer: a Prospective Observational Cohort Study
Brief Title: Association of Sleep Quality and Mental Status With Early Recurrence and Prognosis of Colorectal Cancer
Status: Enrolling by invitation | Type: Observational
Sponsor: Ma Yanlei (Other)
Responsible Party: Sponsor-Investigator, Ma Yanlei, Chief physician, Fudan University
Organization: Fudan University (Other)
Other Study IDs: FDCRC97-MYL
Record Dates: First submitted 2024-05-15; First posted 2024-06-05 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-05

CONDITIONS: Colorectal Cancer; Sleep Quality; Mental Status Change
MeSH Terms: conditions — Colorectal Neoplasms; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective observational cohort study to explore the effects of sleep quality and mental status on early postoperative recurrence and prognosis in patients with colorectal cancer.

DETAILED DESCRIPTION:
Evidence of evidence-based medicine shows that patients with malignant tumors have heavy psychological pressure after disease, and are prone to different degrees of sleep disorders and mental health problems, which often affect the progression and prognosis of the primary tumor. Previous studies have reported that baseline sleep quality was independently associated with risk of progression, risk of death, and response to treatment in patients with metastatic colorectal cancer before and during chemotherapy. Surgery, as a stressor, often causes obvious psychological stress reactions in patients, resulting in varying degrees of sleep disorders and poor mental performance, which may also become a factor affecting the recurrence and prognosis of patients. Therefore, the Department of Colorectal Surgery, Affiliated Cancer Hospital of Fudan University intends to conduct a prospective observational cohort study on the effects of sleep quality and mental state on early postoperative recurrence and prognosis of patients with colorectal cancer, in order to explore the effects of sleep quality and mental state on early postoperative recurrence and prognosis of patients with colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Preoperative fibrocolonoscopy and pathological examination confirmed colorectal cancer;
2. Age 18 ~ 80 years old;
3. Baseline clinical stage TNM Ⅰ to Ⅲ : cT1-4N0-2M0 (AJCC-8 version);
4. The United States Eastern Oncology Consortium (ECOG) physical status score was 0 to 2 points;
5. Laboratory examination results before admission met the following surgical conditions: neutrophil (ANC) ≥1.5×109/L, platelets (PLT) ≥ 100×109/L, total bilirubin (TBI) ≤1.5× upper limit of normal (2mg/dl), alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≤2× upper limit of normal; Coagulation parameters in the normal range;
6. Able to complete the required research questionnaire independently or with the assistance of the researcher;
7. Patients were willing to undergo regular follow-up after surgery and had no psychological, family, social, or geographic constraints that affected protocol compliance and follow-up time;
8. Patients and their families can understand and are willing to participate in this clinical study, and sign informed consent.

Exclusion Criteria:

1. Under 18 years of age or over 80 years of age;
2. Have a family history of severe mental illness;
3. People with mental illness or intellectual disability who cannot correctly describe their feelings;
4. The patient has severe systemic infection;
5. No radical operation was performed during the operation due to various reasons;
6. Patients with intestinal obstruction, intestinal perforation, intestinal bleeding, peritonitis, etc. requiring emergency surgery;
7. Merge other parts of the transfer;
8. Have serious heart, lung, liver and kidney diseases, can not tolerate surgery;
9. Active stage of liver disease or abnormal liver function, ALT, AST, TBIL is more than 2 times the upper limit of normal value;
10. Renal function damage, Cr ≥ 2 times the upper limit of normal value or BUN ≥ 2 times the upper limit of normal value;
11. The subject's blood white blood cells are lower than the lower limit of normal, or platelets are lower than the lower limit of normal, or there are other blood system diseases;
12. Severe coagulation mechanism disorder and bleeding tendency;
13. Serious uncontrolled medical disease, recent history of myocardial infarction (within 3 months); Acute infection;
14. Patients with uncontrolled severe hypertension and severe diabetes after intervention;
15. The researchers considered that other candidates were not suitable for inclusion in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were diagnosed with colorectal cancer by histopathology at the Affiliated Cancer Hospital of Fudan University and underwent surgery for colorectal cancer at the Affiliated Cancer Hospital of Fudan University
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | through study completion, an average of 1 year
  The duration between the date after surgery to the date of any recurrence or death firstly
Overall Survival | through study completion, an average of 1 year
  Time from the start of surgical randomization to death (from any cause)
Effect of sleep quality and mental state on early recurrence and prognosis of patients with colorectal cancer after surgery | through study completion, an average of 1 year
  The correlation of GAD-7 scale score, PHQ-9 scale score and ESAS scale score with Disease-free survival (DFS), Overall Survival and tumor-free survival rate of patients was analyzed

SECONDARY OUTCOMES:
Tumor markers CEA, CA19-9 was used to determine recurrence in patients with colorectal cancer enrolled in the study. | From date of randomization until the date of death from any cause, whichever came first, assessed up to 100 months
  Tumor markers CEA, CA19-9 was used to determine recurrence in patients with colorectal cancer enrolled in the study. 1, 3, 6, 12, 18, 24 months after the operation until the observation endpoint appeared.
Enteroscope was used to determine recurrence in patients with colorectal cancer enrolled in the study. | From date of randomization until the date of death from any cause, whichever came first, assessed up to 100 months
  Enteroscope was used to determine recurrence in patients with colorectal cancer enrolled in the study. 1, 3, 6, 12, 18, 24 months after the operation until the observation endpoint appeared.
Physical examination was used to determine recurrence in patients with colorectal cancer | From date of randomization until the date of death from any cause, whichever came first, assessed up to 100 months
  Physical examination was used to determine recurrence in patients with colorectal cancer.1, 3, 6, 12, 18, 24 months after the operation until the observation endpoint appeared.

CONTACTS AND LOCATIONS:
Overall Officials: Yanlei Ma, PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China